CLINICAL TRIAL: NCT02733757
Title: Effects of Clonidine Added to Lidocaine in Sub-Tenon's and Peribulbar Anesthesia: Assessments of Intraocular Pressure (IOP), Ocular Perfusion Pressure (OPP) and Ocular Pulse Amplitude (OPA)
Brief Title: Clonidine Added Lidocaine in Intraocular Pressure and Hemodynamics Ocular in Sub-Tenon's and Peribulbar Anesthesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Federal University of Espirito Santo (Other)
Responsible Party: Principal Investigator, Renato Santiago Gomez, Head of surgery department of the medical school of the Federal University of Minas Gerais, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAAE - 03409512.2.0000.5149
Record Dates: First submitted 2016-03-15; First posted 2016-04-11 (Estimated); Results first posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Anesthesia
Keywords: Clonidine; Sub-Tenon's and Peribulbar block; IOP; OPP; OPA
MeSH Terms: interventions — Clonidine; Diazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sub-Tenon's group control (No Intervention): 2% Lidocaine without epinephrine
- Sub-Tenon's group clonidine (Experimental): 2% Lidocaine without epinephrine plus clonidine 1 µg/kg
  Interventions: Drug: Clonidine
- Peribulbar group control (No Intervention): 2% Lidocaine without epinephrine
- Peribulbar group clonidine (Experimental): 2% Lidocaine without epinephrine plus clonidine 1 µg/kg
  Interventions: Drug: Clonidine

INTERVENTIONS:
Drug: Clonidine — Clonidine 1 µg/kg plus 2% lidocaine
  Other Names: Atensine
  Arms: Peribulbar group clonidine; Sub-Tenon's group clonidine

SUMMARY:
Regional anesthesia in orbit can reduce ocular blood flow, increase in intraocular pressure (IOP) or the pharmacological action of local anesthetics. This study was conduced to evaluate the effects of clonidine added to lidocaine in IOP, ocular perfusion pressure (PPO) and ocular pulse amplitude (OPA) in patients undergoing cataract surgery under sub-Tenon's and peribulbar anesthesia.

DETAILED DESCRIPTION:
In this prospective randomized and double blind clinical study, involving 80 patients with ages from 30 to 86 years old, ASA I and II, both genders. The patients were randomly divided into 4 groups of 20 patients, and then were administered in control sub-Tenon's group 5 mL of 2% lidocaine with 1 mL of 0.9% sodium chloride solution; in sub-Tenon's group clonidine, 5 mL of 2% lidocaine associated with 1 µg/kg of clonidine diluted in 1 mL 0.9% sodium chloride solution. In the peribulbar anesthesia, the control group with 6 mL of 2% lidocaine and 1 mL of 0.9% sodium chloride solution, and peribulbar group clonidine, 6 mL of 2% lidocaine associated with 1 µg/kg of clonidine diluted in 1 mL 0.9% sodium chloride solution. Were evaluated the systemic hemodynamic variables; IOP and OPA measurements according the dynamic contour tonometer (DCT) and calculation of OPP, prior to the blockade (M0), and one (M1), five (5) and ten minutes (M10) after the injection of the anesthetic solutions. Complications related to the sub-Tenon's and peribulbar anesthesia were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 30 and 86 years old
* Both genders
* Physical status ASA (American Society of Anesthesiologists) I and II
* Cooperative patients undergoing cataract surgery by phacoemulsification

Exclusion Criteria:

* Patients with communication difficulties
* Allergic to any medication protocol
* Chronic therapy with clonidine
* In use of antihypertensive medication
* Diabetes
* Glaucoma
* Previous surgery in the same eye
* Abnormalities in coagulation

Ages: 30 Years to 86 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-05; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sigmar Cabral, PhD, Principal Investigator — Federal University of Espírito Santo, Vitória; Renato Gomez, PhD, Study Director — Federal University of Minas Gerais, Belo Horizonte

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pianka P, Weintraub-Padova H, Lazar M, Geyer O. Effect of sub-Tenon's and peribulbar anesthesia on intraocular pressure and ocular pulse amplitude. J Cataract Refract Surg. 2001 Aug;27(8):1221-6. doi: 10.1016/s0886-3350(01)00797-0. PMID 11524193
- [Background] Watkins R, Beigi B, Yates M, Chang B, Linardos E. Intraocular pressure and pulsatile ocular blood flow after retrobulbar and peribulbar anaesthesia. Br J Ophthalmol. 2001 Jul;85(7):796-8. doi: 10.1136/bjo.85.7.796. PMID 11423451
- [Background] Cabral SA, Carraretto AR, Brocco MC, Abreu Baptista JF, Gomez RS. Effect of clonidine added to lidocaine for sub-Tenon's (episcleral) anesthesia in cataract surgery. J Anesth. 2014 Feb;28(1):70-5. doi: 10.1007/s00540-013-1660-2. PMID 23797624

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sub-Tenon's Group Control | Sub-Tenon's Group Clonidine | Peribulbar Group Control | Peribulbar Group Clonidine
Started | 20 | 20 | 20 | 20
Completed | 20 | 20 | 20 | 20
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sub-Tenon's Group Control | Sub-Tenon's Group Clonidine | Peribulbar Group Control | Peribulbar Group Clonidine | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (12) | 60 (13) | 64 (14) | 62 (12) | 63 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 14 | 12 | 51
  Male | 7 | 8 | 6 | 8 | 29

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP)
Time Frame: Within 10 minutes before the surgery procedure
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Sub-Tenon's Group Control | Sub-Tenon's Group Clonidine | Peribulbar Group Control | Peribulbar Group Clonidine
Number analyzed (Participants) | 20 | 20 | 20 | 20
mmHg | 18 (3) | 16 (4) | 19 (3) | 16 (4)

ADVERSE EVENTS:
Arm/Group | Sub-Tenon's Group Control | Sub-Tenon's Group Clonidine | Peribulbar Group Control | Peribulbar Group Clonidine
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No